CLINICAL TRIAL: NCT02180360
Title: Eight Weeks of Basic Training in Capoeira Increases Flexibility of Beginners in the Sport
Brief Title: Capoeira Training and Flexibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do vale do São Francisco (Other)
Collaborators: University of Pernambuco (Other); Universidade Federal do Rio Grande do Norte (Other)
Responsible Party: Principal Investigator, Sérgio Rodrigues Moreira, Professor (PhD), Universidade Federal do vale do São Francisco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2014-06-27; First posted 2014-07-02 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-06

CONDITIONS: Flexibility; Range of Motion
Keywords: Capoeira training; Range of motion; Flexibility; beginners

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Capoeira training group (Experimental): The Capoeira training was performed during eight weeks, twice a week with duration of 60min each session, divided in 1) initial part: 10min warm-up with activities of low intensity or the "ginga" used in Capoeira; 2) main part: from the Basic Programmed Lesson (40min) and ; 3) final part: Capoeira presentation of 10min. In this last moment, the participants remained in a circle and, in pairs, executed the movements practiced earlier in the sessions. In order to perform the Basic Programmed Lesson, the activities were divided in four stages, composed by "ginga" and other movements: dodging, unbalancing, traumatizing and acrobatic. The volunteers would perform the initial part of the basic lesson (ex. 1st stage) and afterwards, when performing the subsequent part (ex. 2nd stage), would first repeat the 1st basic lesson, with the purpose of continuing the learning process and improving the previous lesson.
  Interventions: Other: Capoeira training group
- Control group (No Intervention): The Control group did not perform any physical exercise during the intervention period (eight weeks).

INTERVENTIONS:
Other: Capoeira training group — Capoeira training: The experimental Capoeira training protocol, based in the modern styles of Capoeira was applied by an instructor with 17 years of experience in teaching Capoeira, followed the directions of the Basic Programmed Lesson, created by Geraldo Pereira d'Santana (Master Santana) in a Capoeira group called IUNA from the city of São Paulo, Brazil.
  In order to perform the Basic Programmed Lesson program, the activities were divided in four stages, being composed of the main movement that characterizes Capoeira (the "ginga") and by other movements such as: dodging, unbalancing, traumatizing and acrobatic.
  An important thing to highlight in the experimental protocol is that the training performed in the present study used only specific movements of Capoeira, without applying any other traditional stretching exercises. Therefore, it is possible to infer that the results obtained are due to the experimental protocol.
  Arms: Capoeira training group

SUMMARY:
Background: Nowadays, a commonly used sport that helps enhancing physical fitness components, including flexibility, is Capoeira. This modality is defined as an athletic sport composed by an individual attack and defensive system, which was originally created in colonial Brazil. Capoeira is characterized by its main movement, the "ginga", and by other several dodging, unbalancing, traumatizing and acrobatic movements. The literature empirically discusses that Capoeira contributes in general physical fitness by modulating several variables of human movement. Among these variables it is possible to highlight the influence of Capoeira in the amplitude of movement of the practitioner's joints. However, no study with a control group has investigated the alterations in flexibility of beginners using an experimental protocol based exclusively in basic techniques of Capoeira, without applying any usual stretching exercises that are commonly used, independently of the specificity of the sport. Objective: To analyze the effects of eight weeks of basic training in Capoeira on the flexibility of beginners in the sport. Methods: Twenty-one individuals, divided in two groups [Capoeira, n=13; 26.1±7.2 years; 22.7±2.7 kg.m2(-1) and Control, n=8; 27.1±0.5 years; 24.3±3.3 kg.m2(-1)] participated in the study. The Capoeira group performed eight weeks of basic training (two sessions per week lasting 60 minutes each). The experimental protocol used was exclusively based in basic techniques of a programmed Capoeira training system. Before and after the intervention measurements were performed aiming to analyze: trunk flexion flexibility, through a sit-and-reach test using a Wells' Bench (WBtf); and passive tension (PThf) and maximum amplitude of hip flexion (MAhf) through goniometry. The hypothesis of this study is that the group Capoeira (beginners) will increase the linear and angular flexibility after eight weeks of basic training in the sport.

ELIGIBILITY:
Inclusion Criteria:

1. All participants had at least a 24 month period without practicing Capoeira;
2. To participate in at least 80% of the experimental sessions (Capoeira group); 4) Not having any kind of bone, muscle or joint impairment that would preclude participating in the study and performing the flexibility evaluations before and after the intervention;
3. Not participating in another physical activity program during the intervention and; 4) Not having any kind of heart disease.

   -

   Exclusion Criteria:

   -

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2012-02; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Trunk flexion flexibility by sit-and-reach test using a Wells' Bench (WBtf - cm); Passive tension (PThf - angle) and Maximum amplitude of hip flexion (MAhf - angle) using goniometry. | Pre-training (Week zero) in Capoeira training group and Control group

SECONDARY OUTCOMES:
Trunk flexion flexibility by sit-and-reach test using a Wells' Bench (WBtf - cm); Passive tension (PThf - angle) and Maximum amplitude of hip flexion (MAhf - angle) using goniometry. | Post-training (after eight weeks) in After eight weeks of Capoeira training group and Control group
Trunk flexion flexibility by sit-and-reach test using a Wells' Bench (WBtf - cm); Passive tension (PThf - angle) and Maximum amplitude of hip flexion (MAhf - angle) using goniometry. | Comparison of pre (0 week) vs. post-training (eight weeks) measures

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio R Moreira, PhD, Principal Investigator — Universidade Federal do vale do São Francisco
Locations (1):
- Universidade Federal do Vale do São Francisco, Petrolina, Pernambuco, Brazil